CLINICAL TRIAL: NCT06818578
Title: Evaluation of the Clinical and Radiographic Success of Different Antibiotic Combinations in Lesion Sterilization and Tissue Repair Therapy for Infected Primary Molar Teeth
Brief Title: Success of Lesion Sterilization and Tissue Repair Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, rüveyda nur culfa, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/74
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Primary Teeth; Pulp Necrosis; Pulpitis - Irreversible
Keywords: lesion sterilization and tissue repair; antibiotics
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Intervention Model Description: This study was a randomized controlled clinical trial that followed the recommendations of the Consolidated Standards of Reporting Trials (CONSORT).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3Mix-MP (Experimental): Metronidazole (Flagyl 500 mg tablets, Sanofi-Aventis, Turkiye), ciprofloxacin (Cipro, 750 mg tablets, Biofarma, Turkiye) and minocycline (Minoz, 100 mg, Ranbaxy, India)
  Interventions: Procedure: Lesion Sterilization and Tissue Repair Therapy; Drug: Different Antibiotic Combinations
- Alternative 3Mix-MP (Active Comparator): Metronidazole (Flagyl 500 mg tablets, Sanofi-Aventis, Turkiye), ciprofloxacin (Cipro, 750 mg tablets, Biofarma, Turkiye) and clindamycin (Klindan, 150 mg capsules, BİLİM, Turkiye)
  Interventions: Procedure: Lesion Sterilization and Tissue Repair Therapy; Drug: Different Antibiotic Combinations

INTERVENTIONS:
Procedure: Lesion Sterilization and Tissue Repair Therapy — LSTR treatment is a minimally invasive, cost-effective, and easy-to-apply procedure for necrotic primary teeth, with a focus on disinfection with an antibiotic mixture without the need for root canal instrumentation.
Drug: Different Antibiotic Combinations — Clinical and Radiographic Success of Different Antibiotic Combinations (evaluating whether the alternative 3Mix-MP combination of clindamycin instead of minocycline is as effective as the standard 3Mix-MP formulation) in Lesion Sterilization and Tissue Repair Therapy
  Other Names: 3Mix-MP and Alternative 3Mix-MP

SUMMARY:
This study aimed to assess the clinical and radiographic success of lesion sterilization and tissue repair (LSTR) therapy with different antibiotic combinations, focusing on evaluating whether the alternative combination of clindamycin instead of minocycline is as effective as the standard 3Mix-MP formulation.

DETAILED DESCRIPTION:
All the clinical procedures were carried out by one clinician with 2 years of clinical experience in pediatric dentistry under rubber dam isolation and local anesthesia via mandibular nerve block. (Maxicaine Fort Ampoule, VEM, Turkiye). After the removal of carious tissues, an endodontic cavity was prepared, and infected coronal pulp tissue was removed up to the canal orifices via a sterile round steel bur. A sterile round steel bur was then used to prepare a medication cavity 2 mm deep and 1 mm wide. The root canals were not instrumented, and only the access cavity was irrigated with a 2.5% NaOCl solution. In cases where hemostasis could not be achieved, a sterile cotton pellet soaked in 5% NaOCl was placed in the pulp chamber and left for 1 minute. Once hemostasis was achieved, the endodontic cavity was dried using a sterile, dry cotton pellet. Pastes were then applied to the medication cavity and covered with a glass ionomer cement (Nova Glass II F, Imicryl, Turkiye) and a stainless steel crown (Kids Crown, Shinhung, Seoul, Korea) at the same visit. Clinical and radiographic evaluations were performed at 1, 3, 6, 9, and 12 months. During follow-up, the teeth were assessed on the basis of the following clinical criteria: pain, dentoalveolar abscess and/or fistula, and tooth loss. The radiographic criterion was periapical radiolucency.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous pain
* Pain on percussion
* The presence of abnormal or pathological mobility
* The presence of a sinus tract or dentoalveolar abscess
* Widening of the periodontal ligament
* Periradicular radiolucency
* Evidence of external and/or internal resorption.

Exclusion Criteria:

* Who required infective endocarditis prophylaxis
* Who had used antibiotics in the two weeks prior to treatment
* İndividuals allergic to the medications used in the study
* Teeth with pulp floor perforation
* Advanced internal and/or external root resorption
* Root canal obliteration
* Excessive bone loss in the furcation area involving the permanent tooth follicle
* Teeth with severe coronal destruction, nonrestorable.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
clinical success | 12 months
  clinical criteria: pain, dentoalveolar abscess and/or fistula, and tooth loss.
radiographic success | 12 months
  radiographic criterion was periapical radiolucency.
overall success | 12 months
  If at least one of the clinical findings was present, the treatment was considered unsuccessful. However, even if teeth fail radiographically, they are not classified as overall failure if no clinical signs are present.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Faculty of dentistry, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided